CLINICAL TRIAL: NCT00376220
Title: A Double-Blind Placebo Controlled Trial of Riluzole in Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-04-23-10
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Drug: Riluzole Initially dispensed 50 mg capsules to take twice a day (BID). At two weeks, increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID (two capsules in the morning (qAM), two capsules in the evening (qHS). If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as Montgomery Asberg Depression Rating Scale (MADRS) < 12) the dose will not be increased further unless clinical symptoms recur.
  Other Names:
  • Rilutek
  Interventions: Drug: Riluzole
- 2 (Placebo Comparator): Initially dispensed 50mg capsules to take BID. At two weeks increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID (two capsules qAM, two capsules qHS). If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as MADRS < 12) the dose will not be increased further unless clinical symptoms recur.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Riluzole — Initially dispensed 50 mg capsules to take twice a day (BID). At two weeks, increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID (two capsules in the morning (qAM), two capsules in the evening (qHS). If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as Montgomery Asberg Depression Rating Scale (MADRS) < 12) the dose will not be increased further unless clinical symptoms recur.
  Other Names: Rilutek
  Arms: 1
Other: Placebo — Initially dispensed 50mg capsules to take BID. At two weeks increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID (two capsules qAM, two capsules qHS). If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as MADRS < 12) the dose will not be increased further unless clinical symptoms recur.
  Arms: 2

SUMMARY:
The Johns Hopkins Department of Psychiatry is conducting a research study to examine the effectiveness of riluzole in treating the depressed phase of bipolar disorder. This outpatient treatment study of medication or placebo will last 9-12 weeks. The study includes medical and psychiatric evaluations as well as time-limited medication treatment at no cost, and you will be compensated for your participation.

DETAILED DESCRIPTION:
The study will last 8 to 12 weeks and requires weekly visits. Participants will come to Johns Hopkins for a screening visit during which they will talk with a psychiatrist, answer questions about their mood and symptoms, have their blood drawn and have a brief physical exam. If they meet criteria for the study, any antidepressant medication that they are taking will be tapered and stopped before beginning study medications. Participation in the study includes free study medication, labs, and testing plus reimbursement for transportation. Participants will also be paid and after the study referred back to their treating psychiatrist with treatment recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* Diagnosed with Bipolar I or II disorder and currently depressed
* Tried at least one antidepressant during the current episode of depression
* Currently taking either lithium, depakote, or tegretol
* Currently in outpatient treatment with a psychiatrist

Exclusion Criteria:

* Current psychotic symptoms
* Women who are pregnant or nursing
* Any serious, uncontrolled medical illness
* History of liver problems
* Current or past blood diseases
* Current drug or alcohol abuse
* Currently receiving Electroconvulsive Shock Therapy (ECT)
* Judged to be at serious suicidal risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2004-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Payne, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zarate CA Jr, Quiroz JA, Singh JB, Denicoff KD, De Jesus G, Luckenbaugh DA, Charney DS, Manji HK. An open-label trial of the glutamate-modulating agent riluzole in combination with lithium for the treatment of bipolar depression. Biol Psychiatry. 2005 Feb 15;57(4):430-2. doi: 10.1016/j.biopsych.2004.11.023. PMID 15705360
- [Background] Zarate CA Jr, Payne JL, Quiroz J, Sporn J, Denicoff KK, Luckenbaugh D, Charney DS, Manji HK. An open-label trial of riluzole in patients with treatment-resistant major depression. Am J Psychiatry. 2004 Jan;161(1):171-4. doi: 10.1176/appi.ajp.161.1.171. PMID 14702270

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment Group: Riluzole: Initially dispensed 50 mg capsules to take twice daily (BID). At two weeks, increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID [two capsules in the morning (qAM), two capsules in the evening (qHS)]. If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as MADRS < 12) the dose will not be increased further unless clinical symptoms recur.
- Inactive/ Placebo Group: Placebo: Initially dispensed 50mg capsules to take BID. At two weeks increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID (two capsules qAM, two capsules qHS). If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as MADRS < 12) the dose will not be increased further unless clinical symptoms recur.
Period: Overall Study
Arm/Group | Active Treatment Group | Inactive/ Placebo Group
Started | 47 | 47
Completed | 37 | 35
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 7 | 10
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Mean age was 43 years old. 58.51 % of the study participants where female and 41.49% were men. The participants were 73% white, non-Hispanic, 21% African-American, non -Hispanic, 4% Latino/Hispanic, and 1% Asian.
Groups:
- Active Treatment Group: Riluzole: Initially dispensed 50 mg capsules to take BID. At two weeks, increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID (two capsules qAM, two capsules qHS). If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as MADRS < 12) the dose will not be increased further unless clinical symptoms recur.
- Inactive/Placebo Group: Placebo: Initially dispensed 50mg capsules to take BID. At two weeks increase dose to 50 mg/100 mg. At four weeks increase to 100 mg BID (two capsules qAM, two capsules qHS). If significant side effects occur (at any time), titration can be slowed and doses can be reduced to a minimum daily dose of 50 mg/day, after which titration may resume by no more than 50 mg a week. Subjects who are unable to tolerate the minimal daily dose permitted in the study will be discontinued from further participation. In addition, if clinical remission is observed at a lower dose of study medication (defined as MADRS < 12) the dose will not be increased further unless clinical symptoms recur.
- Total: Total of all reporting groups
Arm/Group | Active Treatment Group | Inactive/Placebo Group | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 47 | 94
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (10) | 43 (11) | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 43 | 46 | 89
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 33 | 36 | 69
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 94
Montgomery Asberg Depression Rating scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Asberg Depression Rating Scale measures symptoms of depression. The scale is composed of 10 questions with a fixed 7 point scale (0-6). Total score ranges from 0-60. A higher score indicates more depressive symptoms.
  units on a scale | 32.4 (6.7) | 30.4 (6.0) | 31.4 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to the End of 8 Weeks of Therapy.
Description: The Montgomery Asberg Depression Rating Scale measures symptoms of depression (MADRS) is a semi-structured interview rating scale for depression that assesses 10 symptoms. The scale is composed of 10 questions with a fixed 7 point scale (0-6). Total score ranges from 0-60. A higher score indicates more depressive symptoms. MADRS Response will be defined as a > 50% reduction in MADRS score from baseline.
Time Frame: 8 weeks
Population: Discrepancies in number of participants analyzed are due to subjects who dropped out and did not have final assessments. Imputed data was used for those participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment Group | Inactive/Placebo Group
Number analyzed (Participants) | 47 | 47
units on a scale
  Baseline MADRS | 32.4 (1.0) | 30.4 (0.9)
  Week 8 | 21.7 (1.8) | 19.0 (2)

ADVERSE EVENTS:
Arm/Group | Active Treatment Group | Inactive/Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No